CLINICAL TRIAL: NCT03547752
Title: Inmediate Effect of the Visualization of Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OA plus MI in neck pain
Record Dates: First submitted 2018-05-01; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Neck Pain; Chronic Pain; Musculoskeletal Pain
Keywords: motor imaginery; mental training
MeSH Terms: conditions — Neck Pain; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effective movement group (Active Comparator): Observation of a video of neck movement at 100% range of movement, and imagination of the same observed movement, feeling the realization of the movement but not developing it.
  Interventions: Other: observed action and motor imaginery
- Ineffective movement group (Experimental): Observation of a video of neck movement at 40% range of movement, and imagination of the same observed movement, feeling the realization of the movement but not developing it.
  Interventions: Other: observed action and motor imaginery

INTERVENTIONS:
Other: observed action and motor imaginery — Observation of a video of neck movement and imagination of the same observed movement, feeling the realization of the movement but not developing it.

SUMMARY:
The observation of actions and motor imagery has demonstrated the activation of certain mechanisms similar to those that occur during active movement, which could induce immediate changes in the amplitudes of movement and sensorimotor variables in observed and imagined movements. The main aim of the study was test the immediate effect of a protocol of observed actions and motor imagery on cervical range of motion and pain intensity in patients with non-specific chronic neck pain (NSCNP). Randomized double-blind clinical trial in patients with DCCI at a primary health care center in the Community of Madrid. A random distribution of study subjects was made into two groups: a) cervical motion videos were presented at full range of motion and b) the videos presented showed a range of motion limited to 40%. In both groups, visualization tasks of actions were alternated with internal kinesthetic motor imagery, in periods of 1min in 2 consecutive series and with a total of 12 minutes of intervention. Cervical range of motion was assessed with a cervical goniometer and pain intensity immediately following the intervention with an Analog Visual Scale.

ELIGIBILITY:
Inclusion Criteria:

* Nos-Specific Chronic Neck Pain lasting more than 3 months

Exclusion Criteria:

* Systemic Disease diagnosed (i.e. Lupus, Fibrolyalgia or Rheumatoid Arthritis)
* Background of fractures or surgery in the cervical region
* congenital anomalies known
* infectious processes or diagnosis of active cancer at the time of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Cervical Range of Movement | at the beginning and after the intervention, until the end of the study (24 hours)
  CROM goniometer

SECONDARY OUTCOMES:
Cervical Pain Disability | at the beginning and end of the intervention, until the end of the study (24 hours)
  Neck Disability Index
Pain Intensity | at the beginning and end of the intervention, until the end of the study (24 hours)
  Visual Ananlogue Scale: 10cm line, were the left limit means "no pain" and the right limit means "worst imaginable pain"
Catastrophizism | at the beginning and end of the intervention, until the end of the study (24 hours)
  Pain Catastrophizing Scale
Health Related Quality of Life | at the beginning and end of the intervention, until the end of the study (24 hours)
  EuroQoL-5D-5L
Anxiety and Depression | at the beginning and end of the intervention, until the end of the study (24 hours)
  Hospital Anxiety and Depression Scale (HADs)

CONTACTS AND LOCATIONS:
Locations (1):
- CS Entrevías, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Hecke O, Torrance N, Smith BH. Chronic pain epidemiology and its clinical relevance. Br J Anaesth. 2013 Jul;111(1):13-8. doi: 10.1093/bja/aet123. PMID 23794640
- [Background] Munoz-Garcia D, Gil-Martinez A, Lopez-Lopez A, Lopez-de-Uralde-Villanueva I, La Touche R, Fernandez-Carnero J. Chronic Neck Pain and Cervico-Craniofacial Pain Patients Express Similar Levels of Neck Pain-Related Disability, Pain Catastrophizing, and Cervical Range of Motion. Pain Res Treat. 2016;2016:7296032. doi: 10.1155/2016/7296032. Epub 2016 Mar 29. PMID 27119020
- [Background] Niddam DM, Lee SH, Su YT, Chan RC. Brain structural changes in patients with chronic myofascial pain. Eur J Pain. 2017 Jan;21(1):148-158. doi: 10.1002/ejp.911. Epub 2016 Jun 28. PMID 27352085
- [Background] Mao C, Wei L, Zhang Q, Liao X, Yang X, Zhang M. Differences in brain structure in patients with distinct sites of chronic pain: A voxel-based morphometric analysis. Neural Regen Res. 2013 Nov 15;8(32):2981-90. doi: 10.3969/j.issn.1673-5374.2013.32.001. PMID 25206618
- [Background] Eaves DL, Riach M, Holmes PS, Wright DJ. Motor Imagery during Action Observation: A Brief Review of Evidence, Theory and Future Research Opportunities. Front Neurosci. 2016 Nov 21;10:514. doi: 10.3389/fnins.2016.00514. eCollection 2016. PMID 27917103